CLINICAL TRIAL: NCT02285556
Title: The Diagnostic Assessment and Intervention Study of Amphetamine Type Stimulus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Min ZHAO, Vice President, Shanghai Mental Health Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: MZhao-003
Record Dates: First submitted 2014-08-19; First posted 2014-11-07 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Amphetamine Addiction
Keywords: drug carving changes during rehabilitation; community; DNA
MeSH Terms: conditions — Amphetamine-Related Disorders | interventions — Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- general information (No Intervention): use cross-sectional study to collect 1000 ATS abuse or dependence patients' general information and 5 ml blood,get their blood plasma and DNA sample in order to explore the possible addict mechanism.
- ATS diagnosis and evaluation for abusers (No Intervention): Use cohort study design to establish ATS abuse induced craving experiment.Do the initial and follow-up assessment from start smoking to stop smoking after 4 weeks, 12 weeks, 26 weeks, 52 weeks and 26 weeks of returning to the community . Thus compare with normal group to explore the possible psychological abuse mechanism.
- psychological training intervention (Active Comparator): The main content is self-awareness training, social and moral strengthening, impulse control training , problem solving training , situational awareness training , HIV prevention, social skills training under the family atmosphere , family social skills training , interpersonal skills training, community interaction skills training , psychiatric symptoms of self-monitoring skills training and so on.
  Interventions: Behavioral: psychological rehabilitation training
- brain stimulation intervention (Active Comparator): Use randomized, prospective pseudo stimulus controlled clinical trial design, evaluation of repetitive transcranial magnetic stimulation of the left frontal lobe dorsal lateral effect on ATS dependent induced cognitive dysfunction and other symptoms.
  Interventions: Radiation: rTMS 10HZ high frequency stimulation
- ATS diagnosis and evaluation for normal people (No Intervention): Do the same initial and follow-up assessment as ATS abusers who stop smoking after 4 weeks, 12 weeks, 26 weeks, 52 weeks and 26 weeks of returning to the community .
- physical and neurological rehabilitation (Active Comparator): The main content is drug rehabilitation exercise and functional physical training. Rehabilitation led by the discipline cadres , practice once a day, each lasting about 15 minutes .
  Interventions: Behavioral: physical and neurological rehabilitation training
- fake brain stimulation intervention (Placebo Comparator): fake transcranial magnetic stimulation of the left frontal lobe dorsal lateral effect on ATS dependent induced cognitive dysfunction and other symptoms.
  Interventions: Radiation: fake rTMS 10HZ high frequency stimulation

INTERVENTIONS:
Behavioral: psychological rehabilitation training — The main content is self-awareness training, social and moral strengthening, impulse control training , problem solving training , situational awareness training , HIV prevention, social skills training under the family atmosphere , family social skills training , interpersonal skills training, community interaction skills training , psychiatric symptoms of self-monitoring skills training and so on.
  Arms: psychological training intervention
Behavioral: physical and neurological rehabilitation training — The main content is drug rehabilitation exercise and functional physical training. Rehabilitation led by the discipline cadres , practice once a day, each lasting about 15 minutes .
  Arms: physical and neurological rehabilitation
Radiation: rTMS 10HZ high frequency stimulation — Stimulate the dorsolateral prefrontal and parietal lower part , 4 weeks of therapeutic intervention (5 times / week).
  Arms: brain stimulation intervention
Radiation: fake rTMS 10HZ high frequency stimulation — Fake stimulate the dorsolateral prefrontal and parietal lower part , 4 weeks of therapeutic intervention (5 times / week).
  Arms: fake brain stimulation intervention

SUMMARY:
The purpose of this research is to inspire new medical ideas using brain image technology for the treatment of Amphetamine Type Stimulus addition, at the same time lowing the addition damage.

DETAILED DESCRIPTION:
The study will increase the sample size based on the preliminary work,also, establish drug dependence induced craving associated environmental experiments , by using the multi-lead biofeedback instrument , CogState tester, event-related potentials Recorder and 3.0T high-field magnetic resonance imaging system to record the physiology , electrophysiology and brain changes during craving, taking a subjective self-assessment , clinical observations and physiological responses combined system to evaluate the ATS addiction degree.

ELIGIBILITY:
Inclusion Criteria:

* No previous history of any mental disorder meet the DSM-IV diagnosis
* aged 18-49 years old , men and women
* junior high school or higher education
* use of amphetamine-type substances time for more than one year
* cumulative use of amphetamines, substances dose of 50 grams or more.

Exclusion Criteria:

* Current or past had suffered neurological diseases
* exclusion of antisocial personality disorder and borderline personality disorder
* addicts in addition to other substances in tobacco , coffee, social drinking outside
* AIDS virus (HIV) detection positive patients .

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 560 (Actual)
Dates: Start 2012-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
the prevalence of ATS abuse or dependence characteristics and pathogenesis | Baseline
  Plasma and DNA samples were collected to carry out the biochemical genetics and immunology research of ATS abuse or dependence , and to explore the prevalence of ATS abuse or dependence characteristics and pathogenesis.
the physiological psychology and cognitive impairment characteristic of ATS addicts,trends and ATS conducted cases. | Baseline
  Use repeatable battery for the assessment of neuropsychological status(RBANS),Cog-state cognitive function assessment test,event-related potentials(ERPs),functional magnetic resonance imaging(fMRI) in biology ( molecular genetics, blood biochemistry, electrophysiology , imaging ) , psychology, mental health and other aspects of the system to assess the physiological psychology and cognitive impairment characteristic of ATS addicts , trends and ATS conducted cases.

CONTACTS AND LOCATIONS:
Overall Officials: Min Zhao, ph.D., Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China